CLINICAL TRIAL: NCT05225181
Title: Effects of the Combining Physical Exercise and Cognitive Training for the Community-based Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202200014B0
Record Dates: First submitted 2022-01-23; First posted 2022-02-04 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-01

CONDITIONS: Cognitively-normal; Mild Cognitive Impairment; Subjective Cognitive Decline
Keywords: aerobic exercise; cognitive training
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sequential training (Experimental): first perform physical exercise followed by cognitive training
  Interventions: Behavioral: perform physical exercise; Behavioral: cognitive training
- simultaneous training (Experimental): perform physical exercise and cognitive tasks simultaneously
  Interventions: Behavioral: perform physical exercise; Behavioral: cognitive training
- control group (Active Comparator): perform body stretching and health education courses
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: perform physical exercise — one 60-min session of physical training
  Arms: sequential training; simultaneous training
Behavioral: cognitive training — one 60-min session of cognitive training
  Arms: sequential training; simultaneous training
Behavioral: control group — perform body stretching(15min) and health education courses(90min)
  Arms: control group

SUMMARY:
This study aims to (1) determine the intervention effects of sequential and simultaneous training on cognitive function and health-related function for cognitively-normal elderly and elderly with Mild Cognitive Impairment(MCI) and Subjective Cognitive Decline(SCD); (2) compare which combination approach is more advantageous for improvement on outcome measures.

DETAILED DESCRIPTION:
The investigators will recruit 30 cognitively-normal elderly and 30 elderly with Mild Cognitive Impairment(MCI) and 30 elderly with Subjective Cognitive Decline(SCD). Participants will be randomly assigned to one of three groups: sequential training (first perform physical exercise followed by cognitive training), simultaneous training (perform physical exercise and cognitive tasks simultaneously), and control group (perform body stretching and health education courses). All participants will receive trainings for 120 minutes per day, one day per week for 12 weeks. The outcome will include measurements that evaluate the cognitive, physical, daily functions, quality of life, and social participation. Participants will be assessed at baseline, after the intervention, and at 3-month follow-up. Repeated measures of analysis of variance (ANOVA) will be used to evaluate the changes in outcome measures at three different time points for the elderly with cognitively-normal, Mild Cognitive Impairment(MCI) and Subjective Cognitive Decline(SCD), respectively. The investigators also use the analysis of covariance (ANCOVA) to investigate the differences between the Mild Cognitive Impairment(MCI) and Subjective Cognitive Decline(SCD) groups on the outcome measures.

ELIGIBILITY:
cognitively-normal elderly

Inclusion Criteria:

1. age≥60
2. able to follow instruction
3. MoCA>26
4. not SCD or MCI or Dementia

Exclusion Criteria:

1. concomitant neurological conditions such as dementia, Parkinson's disease, brain tumor, brain injury and other brain diseases (such as intracranial hypertension or cerebral edema);
2. have unstable cardiovascular status such as uncontrolled hypertension

SCD

Inclusion Criteria:

1. age>=60
2. SCD(from Ecog-12)
3. MoCA≥26
4. not MCI or Dementia

Exclusion Criteria:

1. concomitant neurological conditions such as dementia, Parkinson's disease, brain tumor, brain injury and other brain diseases (such as intracranial hypertension or cerebral edema);
2. have unstable cardiovascular status such as uncontrolled hypertension

MCI

Inclusion Criteria:

(1)age>=60 (2)20 ≦MoCA < 26 (3)MCI (3)not Dementia

Exclusion Criteria:

1. concomitant neurological conditions such as dementia, Parkinson's disease, brain tumor, brain injury and other brain diseases (such as intracranial hypertension or cerebral edema);
2. have unstable cardiovascular status such as uncontrolled hypertension

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change scores of the Montreal Cognitive Assessment (MoCA). | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Montreal Cognitive Assessment (MoCA) will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitive functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke. The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Wechsler Memory Scale (WMS) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  including Faces Recognition (total scale=48), Verbal Paired Associates (total scale = 32), Word Lists (total scale = 48), and Spatial Span (total scale=32) will be used to assess the immediate, delayed, and working memory tests. For each subtest, a higher number indicates better performance in memory function. The raw score of subtests will also be transferred to standardized Z scores and summed to represent an index of general memory function.
Change scores of Stroop test | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The participants will be tested under congruent and incongruent conditions. In the congruent condition, the participant will name the color ink of a word which is consistent with the written color name; whereas in the incongruent condition the participant will name the color ink differs from the written color name. The time to complete the task will be calculated for each condition
Change scores of Color trials test | baseline, after the intervention eight weeks, and at 3-month follow-up.
  For Part 1, the respondent uses a pencil to rapidly connect circles numbered 1-25 in sequence. For Part 2, the respondent rapidly connects numbered circles in sequence, but alternates between pink and yellow. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors.

SECONDARY OUTCOMES:
Change scores of Verbal fluency tests | baseline, after the intervention eight weeks, and at 3-month follow-up.
  Verbal fluency tests are a kind of psychological test in which participants have to produce as many words as possible from a category in a given time (usually 60 seconds).
Change scores of Wechsler Adult Intelligence Scale; WAIS | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The digit symbol test involves a key consisting of the numbers 1-9, each paired with a unique, easy-to-draw symbol such as a "V", "+" or ">".
  Matrix Reasoning
  This is a nonverbal reasoning task in which individuals are asked to identify patterns in designs. This subtest measures:
  * non-verbal reasoning skills
  * broad visual intelligence
  * perceptual organization skills
Change scores of the short (12-item) form of the Everyday Cognition Scale (ECog-12) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The short (12-item) form of the Everyday Cognition Scale (ECog-12), which was developed as an informant-rated report of cognitively mediated functional abilities in older adults. The ECog-12 asks participants to rate their current ability to perform cognitively mediated daily tasks related to everyday memory, language, visuospatial abilities, and executive functions compared with their ability to do the same task 10 years ago. Items are rated on a scale of 1-4, with 1 = Better or no change and 4 = Consistently much worse. The global, executive, and memory ECog-12 sub-domain scores were generated by averaging over the component items (sum of items/number of items) to maintain a range of 1 to 4 (with higher scores reflecting greater self-reported SCD).
Change scores of Dual-task tests | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The dual-task test evaluates the ability to shift attention between one task and another. Participants will sit and perform the box and block test (BBT) or walk 10 meters while doing secondary cognitive or motor tasks. Two cognitive secondary tasks will be performed by the participants: (1) arithmetic task: participants will be asked to perform serial subtractions by 7 starting from 100 or random two-digit numbers (e.g., Baetens et al., 2013); (2) tone discrimination task: participants will be presented a number of low and high-pitched tones and they will respond to either the high or low-pitched tones during the trial. Both cognitive task performances will be recorded and the results will be compared to single cognitive task performance. In addition to the cognitive dual-task, participants will perform a motor task (e.g., holding a cup of water) while walking.
Change scores of Six-minute walk test,6MWT | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. T
Change scores of Timed up and go (TUG) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The TUG assesses the dynamic balance ability and mobility. The participants will be required to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The time to complete the TUG test has been shown to be a good indicator to detect potential fallers in frail elderly (Podsiadlo & Richardson, 1991). The test-retest reliability of TUG on individuals with cognitive impairment was excellent (Blankevoort, van Heuvelen, & Scherder, 2013).
Change scores of 30 second chair stand test,CST | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The 30 second sit-to-stand will be assessed to indicate the strength and endurance level of the lower extremities. The participants will be asked to stand up from a standardized chair and then sit down as many times as possible within 30 seconds. The feasibility and reliability of using sit-to-stand test in people with cognitive impairment have been established to be good (Blankevoort et al., 2013).
Change scores of International Physical Activity Questionnaires (IPAQ) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Chinese version of the International Physical Activity Questionnaires (IPAQ) is an international measure for health-related physical activity. A short form of IPAQ will be used to assess changes in physical activity before and after intervention in this study. The reliability and validity of IPAQ has been established across 12 countries .
  The self-report, short-form IPAQ , consists of three questions about days and time of vigorous, moderate, and walking activity in bouts of 10 min, with one question about daily sedentary time in the preceding seven days. The questionnaire was preceded by completion instructions and three questions about the types of vigorous, moderate, and light activity undertaken .
Change scores of Grip strength | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The investigator will use hand dynamometer to measure grip strength of both hands while the participant is seated, with the elbow at 90-degree flexion. The investigator will record the mean value of 3 attempts.
  Grip strength was measured using a digital dynamometers method, which is a tool with an adjustable grip span, ranging from 3.5 to 7 cm and weighing from 5 to 100 kg with minimal difference around 0.1 kg . All the participants were in a sitting position with fully extended elbows . Then, the investigator measured Grip strength on the dominant hand after 2-3 minutes of resting.
Change scores of short physical performance battery,SPPB | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older persons. The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests . It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.
Change scores of The Clinical Frailty Scale (CFS) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The aim of this scoping review is to identify and document the nature and extent of research evidence related to the Clinical Frailty Scale (CFS). The association of Clinical Frailty Scale (CFS) score with clinical outcomes highlights its utility in the care of the aging population.
  The Clinical Frailty Scale (CFS) is a judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).
Change scores of Reported Edmonton Frail Scale (REFS) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  Reported Edmonton Frail Scale is an adaptation of Edmonton Frail Scale, that can be performed in less than 10 min by any healthcare professional. Reported Edmonton Frail Scale substitutes the last domain on Edmonton Frail Scale, the physical performance measure, with three self-assessed physical performance questions . This is ideal for use in busy cardiology clinics when patients are being assessed for suitability for intervention.Scoring for the Reported Edmonton Frail Scale range is 0 to18. Not Frail：0-5 ;Apparently Vulnerable：6-7; Mildly Frail：8-9;Moderate Frailty：10-11;Sever Frailty：12-18.
Change scores of Amsterdam Instrumental Activity of Daily Living,A-IADL | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Amsterdam Instrumental Activity of Daily Living (A-IADL) is an adaptive and computerized questionnaire designed to assess impairments in instrumental activities of daily living (IADL) in (early) dementia. The questionnaire is completed by a caregiver, such as a relative or friend.
  Each item has a 5-point scale response option (scored 0-4). The scoring of the Amsterdam Instrumental Activity of Daily Living is calculated using item response theory .Lower scores indicating poorer performance.
Change scores of the World Health Organization Quality of Life-Old(WHOQOL-OLD) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The World Health Organization Quality of Life-Old questionnaires demonstrate acceptable psychometric performance in a convenience sample of Taiwan older people. It are valuable measures of Quality of Life-Old for use with older people.Time frame for assessment is the past two weeks.
  The items are distributed into 4 domains (physical; psychological, social and environmental health) and 25 facets.
Change scores of Geriatric Depression Scale,GDS | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Geriatric Depression Scale (GDS) is a screening test originally developed by J.A. Yesavage and colleagues in 1982 that is used to identify symptoms of depression in older adults. The scale is a 30-item, self-report instrument that uses a "Yes/No" format.
Change scores of Community Integration Questionnaire, CIQ | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The community integration questionnaire (CIQ) was designed to assess home integration, social integration and productive activity in persons with acquired brain injury. The instrument consists of 15 items and can be completed by self report or with the assistance of a family member or caregiver familiar with the person's health status and social activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memotial Hospital, Taoyuan District, Taiwan